CLINICAL TRIAL: NCT02300935
Title: Phase I Study of Trametinib and Nab-paclitaxel in Patients With Melanoma
Brief Title: Study of Trametinib and Nab-paclitaxel in Patients With Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study concept was terminated.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MEL 40
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Melanoma
Keywords: trametinib; nab-paclitaxel; Mekinist; Abraxane; unresectable; metastatic
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — trametinib; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- trametinib and nab-paclitaxel (Experimental): Trametinib will be dosed at 1mg, 1.5mg, and 2mg orally (PO) daily based on Phase I data of this drug as a single agent. All patients entering this study will receive intravenous (IV) nab-paclitaxel on Day 1, 8, and 15. Dose levels will be assigned to each patient, and dose escalation decisions will be based on the evaluation of safety data from the prior cohort.
  Interventions: Drug: trametinib; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: trametinib
  Other Names: Mekinist
Drug: nab-paclitaxel
  Other Names: Abraxane

SUMMARY:
This study will investigate the combination of two drugs, trametinib and nab-paclitaxel, in patients with advanced unresectable or metastatic melanoma. Each drug has shown activity in trials of patients with melanoma. However, the combination of these two drugs has not been studied. In this trial the investigators will determine the maximum dose of the drug combination to be administered to patients with advanced unresectable or metastatic melanoma and examine the safety profile of the drug combination.

DETAILED DESCRIPTION:
While treatment for melanoma has evolved in the last few years, advanced/metastatic melanoma remains an aggressive disease with poor prognosis. Trametinib and nab-paclitaxel have demonstrated single-agent activity in Phase III trials of patients with melanoma. The investigators propose to investigate this drug combination in patients with advanced unresectable or metastatic melanoma. This open-label Phase I study is designed to determine the maximum tolerated dose (MTD), recommended Phase II dose (RP2D), and safety profile of trametinib and nab-paclitaxel given in combination. Patients with melanoma and known BRAF mutation status will receive escalating doses of trametinib and nab-paclitaxel to determine the MTD. Once the MTD is determined an additional 6 patients will be treated at the MTD to establish the dose for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with histologically or cytologically-confirmed advanced unresectable or metastatic melanoma. BRAF mutation-positive and wild-type tumors are allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, renal, and hepatic function
* Life expectancy ≥12 weeks
* Any pre-existing neuropathy must be <grade 2 per Common Technology Criteria for Adverse Events (CTCAE) version 4.0

Exclusion Criteria:

* More than 1 prior cytotoxic chemotherapy regimen in the metastatic setting
* Prior MEK inhibitor therapy (prior BRAF inhibitor allowed)
* Prior nab-paclitaxel (prior taxane allowed)
* Use of an investigational anti-cancer drug within 21 days or 5 half-lives (whichever is shorter) prior to first dose. A minimum of 10 days after termination of investigational drug is required. Any drug-related toxicity should have resolved to Grade 1 or baseline.
* Symptomatic or untreated brain metastases
* History of retinal vein occlusion (RVO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Estimated); Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AEs) as a Measure of Safety and Tolerability | weekly for the first 4 weeks
  The maximum tolerated dose (MTD) of the drug combination will be determined as the highest dose at which ≤1 of 6 patients experience a dose limiting toxicity (DLT) during one cycle (28 days) of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R. Infante, MD, Study Chair — SCRI Development Innovations, LLC
Locations (3):
- United States (3):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Center, Sarasota, Florida
  - Tennessee Oncology PLLC, Nashville, Tennessee